CLINICAL TRIAL: NCT00698438
Title: Prospective, Randomized Clinical Trial,to Compare Standard Trabeculectomy to the Ex-PRESS Mini Glaucoma Shunt Implantation Under a Scleral Flap in Eyes With Open-Angle Glaucoma
Brief Title: Comparison Of Trabeculectomy Versus The Ex-PRESS Miniature Glaucoma Device In The Same Patient: A Prospective Randomized Study
Acronym: XVT-USF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Elie Dahan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XVT-USF
Record Dates: First submitted 2008-03-04; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Glaucoma
Keywords: At least 18 years of age; Open-angle glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a (Active Comparator): Implantation of Ex-PRESS mini glaucoma shunt under a scleral flap
  Interventions: Device: Ex-PRESS implantation; Procedure: Trabeculectomy
- b (Active Comparator): Trabecolectomy
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Device: Ex-PRESS implantation — I. Mobility check of the device. II. Administration of a local or topical anesthetic. III. Preparation and coverage of the eye by conventional sterile procedures. IV. Injection of viscoelastic material into the AC through a paracenthesis. V. Creation of a scleral tunnel up to clear cornea. VI. Creation of a (5 mm) conjunctival tunnel fornix based. VII. Lifting of the conjunctiva and tenon. VIII. Formation of a 2mm scleral incision at 0.3mm depth, 1.5mm from the limbus. IX. Application of 0.5µg/ml MMC under the tunnel for one minute.
  X. Penetration into the AC using a 0.65mm stiletto, inside the tunnel of the sclera-corneal junction.
  XI. Implantation of the Ex-PRESSTM through that pre-incision at the sclerocorneal junction.
  XII. Introducer withdrawal. XIII. Tucking the plate under the scleral tunnel, and verification of the position inside the tunnel.
  XIV. Reposition the conjunctiva with 1 - 2 sutures at the limbus. XV. Closing the conjunctiva with a suture.
  Other Names: a:Ex-PRESS implantation
  Arms: a
Procedure: Trabeculectomy — standard trabeculectomy

SUMMARY:
the purpose of this study was to compare standard trabeculectomy to the Ex-PRESS mini glaucoma shunt implantation under a scleral flap in eyes with open-angle glaucoma.In this report, we describe the results of a prospective, randomized trial in which subjects with bilateral primary open-angle glaucoma underwent the two procedures in fellow eyes.Design: Prospective, randomized clinical trial.

Participants: 15 subjects with bilateral primary open-angle glaucoma Methods: Subjects underwent the two procedures in fellow eyes. Safety and efficacy were evaluated for up to two years.

Main Outcome Measures: Mean IOP and surgical success rates. Results: Mean IOP was similar in Ex-PRESS and trabeculectomy eyes at all time points except month 9, when Ex-PRESS eyes had lower mean IOP (13.2 mmHg vs 16.5 mmHg, respectively; p=0.025). Percent IOP reduction was also similar at all time points except postoperative day 1, when trabeculectomy eyes were lower (75.5% vs 65.8%, respectively; p=0.003), likely due to a higher rate of early hypotony in trabeculectomy eyes versus Ex-PRESS eyes (47% vs 7%, respectively). Complete (without medications) and qualified (with or without medications) successes were more common at all IOP cut-off values in Ex-PRESS eyes than trabeculectomy eyes at last visit (p=0.015, p=0.015 respectively). Postoperative complications were uncommon in both groups, but trabeculectomy eyes required more postoperative interventions than Ex-PRESS eyes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were at least 18 years of age and
* Had medically uncontrolled primary open-angle glaucoma requiring incisional surgery for reduction of intraocular pressure in both eyes.
* Subjects with prior cataract or failed filtration surgery in either eye were eligible to participate if surgery occurred at least 3 months prior to enrollment.

Exclusion Criteria:

* Any form of glaucoma other than primary open-angle glaucoma;
* History of or active uveitis; or
* Any ocular abnormality that would prevent accurate assessment of intraocular pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-03; Primary Completion 2007-08

PRIMARY OUTCOMES:
Mean IOP and surgical success rates. na

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, University of the Witwatersrand,, Johannesburg, South Africa

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740